CLINICAL TRIAL: NCT00183066
Title: Collection of Bone Marrow Aspirate From Volunteer Donors for In Vitro Hematopoietic Research
Brief Title: Collection of Bone Marrow Aspirate From Volunteer Donors
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: AG0046
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Aging

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow aspirates Whole blood

SUMMARY:
The purpose of this study is to collect bone marrow cells for research purposes.

DETAILED DESCRIPTION:
This study is designed to provide bone marrow cells for other research studies. The research is being done because there are ongoing experiments in a number of National Institute on Aging (NIA) laboratories that require access to normal human bone marrow aspirate for their studies of the immune system. These studies are done to understand how blood cells are formed and how they function. Samples will be used to study problems such as the immune system in bone marrow failure and related conditions. Cells will be used in laboratory research and may be banked for future laboratory studies

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers age 18 and over

Exclusion Criteria:

* Significant abnormalities on health history questionnaire or in the results of blood tests
* Pregnant or nursing mother
* Participation in another research study within the past six weeks that is felt by the Principal Investigator to be incompatible with this study
* Severe infection in the past two months
* Immune disorder, or use of any medication that can alter immune system function
* A medical or mental health finding showing inability to go through the procedure
* Body mass index (BMI) greater than 29%
* Chronic back pain, sciatica, or a compression fracture of the spine
* Positive test results for viral infections: Hepatitis B, Hepatitis C, or HIV (AIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy males and females 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2002-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan L. Longo, MD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- NIA Clinical Research Unit located at Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cashman J, Clark-Lewis I, Eaves A, Eaves C. Stromal-derived factor 1 inhibits the cycling of very primitive human hematopoietic cells in vitro and in NOD/SCID mice. Blood. 2002 Feb 1;99(3):792-9. doi: 10.1182/blood.v99.3.792. PMID 11806978
- [Background] Exley MA, Tahir SM, Cheng O, Shaulov A, Joyce R, Avigan D, Sackstein R, Balk SP. A major fraction of human bone marrow lymphocytes are Th2-like CD1d-reactive T cells that can suppress mixed lymphocyte responses. J Immunol. 2001 Nov 15;167(10):5531-4. doi: 10.4049/jimmunol.167.10.5531. PMID 11698421
- [Background] Johnson BS, Mueller L, Si J, Collins SJ. The cytokines IL-3 and GM-CSF regulate the transcriptional activity of retinoic acid receptors in different in vitro models of myeloid differentiation. Blood. 2002 Feb 1;99(3):746-53. doi: 10.1182/blood.v99.3.746. PMID 11806973